CLINICAL TRIAL: NCT06879197
Title: Clinical Relevance of the Major Pathologic Regression for Locally Advanced Rectal Cancer Following Neoadjuvant Chemoradiotherapy: A Multi-center Study
Brief Title: Clinical Relevance of Major Pathologic Regression for Locally Advanced Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, M.D., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: GIH-SYSUyip33
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Rectal Neoplasms; Chemotherapy Effect
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We evaluated all related clinical and pathologic data of patients with Locally Advanced Rectal Cancer following Neoadjuvant Chemoradiotherapy, including the pathologic regression grading, and other histopathologic characteristics. Finally, the present study was aimed at (1) clarifying the clinical significance of the Major Pathologic Regression for Locally Advanced Rectal Cancer following Locally Advanced Rectal Cancer and (2) comparing different Neoadjuvant Chemoradiotherapy treatments of this uncommon disease through conducting a large, multi-center cohort study.

DETAILED DESCRIPTION:
This large-scale, multi-center cohort study aims to investigate the clinical and prognostic implications of histopathologic characteristics in patients with Locally Advanced Rectal Cancer (LARC) following Neoadjuvant Chemoradiotherapy (NCRT). The study will retrospectively and prospectively analyze data from consecutive LARC patients treated at participating institutions between 2016 and 2022.

Study Design and Objectives

Primary Objective:

To evaluate the clinical significance of Major Pathologic Regression (MPR) in LARC patients following NCRT. MPR is defined as ≤10% residual viable tumor within the tumor bed in the pathologic evaluation. The study will correlate MPR status with long-term survival outcomes, including Progression-Free Survival (PFS) and Overall Survival (OS), to determine its validity as a surrogate endpoint for treatment efficacy.

Secondary Objectives:

To compare the efficacy of different NCRT regimens (e.g., fluoropyrimidine-based vs. oxaliplatin-containing protocols) in achieving MPR and improving survival outcomes.

To assess the prognostic value of novel histopathologic parameters, such as tumor necrosis density (NECR-TD), tumor-infiltrating lymphocyte (TLS) density, and TLS-to-necrosis ratio (T/NR), in predicting DFS and OS.

Study Population

Inclusion Criteria:

Adults (≥18 years) diagnosed with locally advanced rectal adenocarcinoma (clinical stage II-III).

Completion of NCRT followed by curative-intent surgery. Availability of pre- and post-treatment histopathologic data, including standardized regression grading and digitized whole-slide images (WSIs).

Exclusion Criteria:

Metastatic disease at diagnosis. Incomplete clinical or pathologic records. Data Collection and Variables

Clinical Data:

Demographics, tumor stage ( ypTNM), NCRT regimen, surgical approach, recurrence, and survival outcomes.

Pathologic Data:

Regression Grading: Residual viable tumor percentage, necrosis extent, and lymph node regression (ypN-Reg+/-).

Quantitative Digital Pathology: AI-driven analysis of WSIs to compute NECR-TD, TLS-TD, and T/NR (Figure 1).

Follow-Up:

PFS and OS will be tracked for a minimum of 3 years post-surgery. Statistical Analysis

Survival Analysis:

Kaplan-Meier curves and Cox proportional hazards models will assess associations between MPR, histopathologic parameters, and survival outcomes.

Comparative Analysis:

Subgroup analyses will compare outcomes across NCRT regimens and LARC subtypes (e.g., mucinous vs. adenocarcinoma).

Machine Learning:

Prognostic models integrating clinical and histopathologic variables will be developed to predict DFS/OS.

Ethical Considerations The Institutional Review Boards (IRBs) of all participating centers have approved the study protocol.

Patient data will be anonymized, and informed consent will be waived for retrospective cohorts but obtained prospectively.

Innovation and Impact

This study addresses critical gaps in the prognostication of LARC by:

Validating MPR as a standardized endpoint for NCRT efficacy. Introducing quantitative, AI-driven histopathologic biomarkers (e.g., T/NR) to refine risk stratification.

Providing evidence for optimizing NCRT regimens based on tumor biology and regression patterns.

Results will be disseminated through peer-reviewed publications and clinical guidelines to improve personalized treatment strategies for LARC.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) diagnosed with locally advanced rectal adenocarcinoma (clinical stage II-III).

Completion of NCRT followed by curative-intent surgery. Availability of pre- and post-treatment histopathologic data, including standardized regression grading and digitized whole-slide images (WSIs).

Exclusion Criteria:

* Metastatic disease at diagnosis. Incomplete clinical or pathologic records.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Locally Advanced Rectal Cancer following Locally Advanced Rectal Cancer
Sampling Method: Probability Sample
Enrollment: 1187 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
PFS | 5 year
  Progression free regression
OS | 5 year
  overall survival